CLINICAL TRIAL: NCT06172413
Title: Twice-daily 15 mA Transcranial Alternating Current Stimulation for Treatment-Resistant Depression
Brief Title: Transcranial Alternating Current Stimulation for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Ningcheng Center Hospital (Unknown); Changning Mental Health Center (Unknown); Tianjin Anding Hospital (Other); Kangning Hospital, Ningbo University (Unknown)
Responsible Party: Principal Investigator, wanghongxing, Professor, MD & PhD, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRD-tACS
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Treatment-Resistant Depression
Keywords: Treatment-Resistant Depression; tACS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active transcranial alternating current stimulation (tACS) (Experimental): true stimulation.
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Sham tACS (Sham Comparator): no active stimulation
  Interventions: Device: Sham tACS

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — Three conductive electrodes will be applied to the scalp: one 4.45 × 9.53 cm electrode placed over the forehead (Fpz, Fp1, and Fp2 in the 10/20 international placement system) and two 3.18 × 3.81 cm electrodes over the mastoid areas.
  The tACS stimulation waveform includes ramp-up and ramp-down periods of 180 and 12 s, respectively. It is a square-wave with an average amplitude of 15 mA and is equally distributed from the frontal region to the mastoid areas (amplitudes are reported as zero-to-peak).
  Each subject will receive 40 sessions of tACS intervention during 4 consecutive weeks at a fixed day time twice per day (once in morning and afternoon, respectively) from Monday through Friday. Each session lasts 40 min.
  Arms: active transcranial alternating current stimulation (tACS)
Device: Sham tACS — Sham tACS
  Arms: Sham tACS

SUMMARY:
This trial aims to investigate the effect of twice-daily 15 mA transcranial alternating current stimulation (tACS) through three conductive electrodes attached to the scalp in subjects with treatment-resistant depression (TRD). Two hundred adult subjects with TRD will be included in this randomized, double-blind, parallelized, multi-centre study. The primary outcome is the change of the Montgomery-Asberg Depression Rating Scale (MADRS) after four weeks of tACS.

DETAILED DESCRIPTION:
This is an 8-week, multicenter, double-blind, sham-controlled, randomized, parallel-group trial.

TRD is defined as failure of response to at least two antidepressant medication trials based on the Massachusetts General Hospital antidepressant treatment response questionnaire (MGH-ATRQ). Patients will be randomized if they remain moderately ill, assessed by Hamilton Depression Scale-item 17 (HAMD-17) score ≥ 20. The primary outcome is a change in the MADRS total score after four weeks of tACS.

"Remission" is defined as MADRS total score ≤10 at Week 4 and Week 8. "Response" is a ≥50% reduction in MADRS total score from baseline to Week 4 and Week 8.

All participants will receive 40 sessions with stimulation at 77.5 Hz and 15 mA (Active group) or sham stimulation (Sham group).

Each session will last 40 minutes from Monday to Friday at a fixed daytime interval for four continuous weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old;
2. able to provide written informed consent;
3. had a diagnosis of major depression disorder (MDD) (recurrent episodes) without psychotic features in compliance with the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revised (DSM-IV-TR) and confirmed by the Mini-International Neuropsychiatric Interview Chinese version 5.0;
4. failure to respond to at least two antidepressant medication trials based on the MGH-ATRQ;
5. ongoing antidepressant(s) at a fixed dose for at least four weeks before baseline assessment;
6. scored≥20 on the Hamilton Depression Scale-item 17 (HAMD-17) at baseline.

Exclusion Criteria:

1. Axis I psychiatric disorders, including schizophrenia, bipolar disorder, manic episodes, anxiety disorders (panic disorder, generalized anxiety disorder, and social anxiety disorder), post-traumatic stress disorder, obsessive-compulsive disorder, anorexia nervosa, bulimia nervosa, psychosis over the previous six months, and any disorders in Axis II (borderline personality disorder, antisocial personality disorder, schizotypal personality disorder, and narcissistic personality disorder);
2. a treatment history of electroconvulsive therapy (ECT), modified ECT, transcranial direct current stimulation, tACS, deep brain stimulation, and transcranial magnetic stimulation (TMS);
3. risk for suicide (defined as a score of ≥ 3 on the suicide item of HAMD-17);
4. known allergy to electrode materials;
5. inability to communicate with researchers fluently;
6. traumatic brain injury;
7. cerebrovascular or cardiovascular stents;
8. substance use disorder (abuse or dependence, as defined by DSM-IV-TR) in the previous six months;
9. for females, pregnant or breastfeeding, or females of childbearing potential refused to use reliable contraceptive methods during the study;
10. dementia (as defined by Short Blessed > 10 and/or clinical evidence of dementia);
11. participated in other clinical research within three months before enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS): Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score After 4 weeks of Treatment | week 0, 4
  The MADRS has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS): remission (defined as MADRS total score ≤10) at Week 4 and Week 8; response is a ≥50% reduction in MADRS total score from baseline to Week 4 and Week 8 | week 0, 4, 8
  The MADRS has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Hamilton Depression Rating Scale (HAMD-17): the changes of HAMD-17 scores and its subscales from baseline to Week 4 and Week 8. | week 0, 4, 8
  HAMD-17 ranges from 0 to 52, with higher scores indicating more depression; a score of 20 or more indicates a moderate to severe depression.
Clinical Global Impression-Severity (CGI-S): the change from baseline to Week 4 and Week 8 in Clinical Global Impression- Severity (CGI-S) | week 0, 4, 8
  The clinical global impression-severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. Score 1 presents normal, not at all ill, and score 7 presents among the most extremely ill patients.
Clinical Global Impression-Improvement (CGI-I): CGI-I score at Week 4 and Week 8. | week 4, 8
  The clinical global impression-improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Score 1 presents the patient as much improved, and score 7 presents much worse.
EuroQol-5 Dimension-level Scale (EQ-5D-5L): the change from baseline to Week 4 and Week 8 in EQ-5D-5L. | week 0, 4, 8
  EQ-5D-5L is an instrument which evaluates the generic quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The score ranges from 5 (having no problems) to 25 (being unable to do/having extreme problems).

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Wang, MD & PhD, Principal Investigator — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao W, Wang H, Leng H, Xue Q, Peng M, Jin X, Tan L, Pan N, Wang X, Wang J, Gao K, Zhang X, Wang H. Acute effect of twice-daily 15 mA transcranial alternating current stimulation on treatment-resistant depression: a case series study. Gen Psychiatr. 2023 Nov 10;36(6):e101278. doi: 10.1136/gpsych-2023-101278. eCollection 2023. No abstract available. PMID 38028814
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/38028814/